CLINICAL TRIAL: NCT03634332
Title: Phase II Study of PEGPH20 and Pembrolizumab (MK-3475) for Patients With Previously Treated Hyaluronan High (HA-High) Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Second-line Study of PEGPH20 and Pembro for HA High Metastatic PDAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pancreatic Cancer Research Team (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Halozyme Therapeutics (Industry); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT 16-001
Record Dates: First submitted 2018-07-23; First posted 2018-08-16 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Pancreatic Neoplasms
Keywords: pancreatic; pancreas; cancer; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Adenocarcinoma | interventions — PEGPH20; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single Treatment Arm for Second-Line treatment of Specific sub-set (HA high) of advanced pancreatic cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PEGPH20 plus Pembrolizumab (Experimental): All patients will receive treatment with PEGPH20 3 micrograms/kg IV weekly x 3, and pembrolizumab 200 mg IV every 3 weeks, in 3-week cycles.
  Interventions: Drug: PEGPH20; Biological: Pembrolizumab

INTERVENTIONS:
Drug: PEGPH20 — PEGPH20 is a PEGylated, neutral-pH-active human hyaluronidase PH20 produced by recombinant DNA technology
Biological: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2
  Other Names: Keytruda; MK-3475

SUMMARY:
This study is the study of the combination of PEGPH20 and Pembrolizumab (MK-3475) for patients with previously treated Hyaluronan High (HA-high) metastatic pancreatic ductal adenocarcinoma. This study is an interventional, unblinded, open label study. Approximately 35 subjects will be enrolled. The trial will require approximately a total of 18 months, including 12 months for enrollment, with an additional 6 months for patient follow-up, data collection and study closure.

Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of up to 21 days, eligible subjects will receive PEGPH20 beginning with Cycle 1 Day 1, on Days 1, 8 15 of every 3 week-cycles and pembrolizumab beginning on Cycle 1 Day 1 (2-4 hrs after PEGPH20), every 3-week-cycles.

Treatment with PEGPH20 and pembrolizumab will continue until progressive disease (PD), unacceptable adverse events (AEs), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, subject receives 35 treatments (approximately 24 months) of pembrolizumab, or administrative reasons requiring cessation of treatment. Subjects who discontinue for reasons other than PD will have post-treatment follow-up for disease status until PD, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival (OS) until death, withdrawal of consent, or the end of the study.

After the end of treatment, each subject will be followed for 30 days for AE monitoring. Serious adverse events (SAE) and events of clinical interest (ECI) will be collected for 90 days after the end of treatment or for 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier.

DETAILED DESCRIPTION:
Combination strategies geared towards blocking the PD1/PD-L1 inhibitory pathway, such as with pembrolizumab, concurrent with stroma depletion (PEGPH20) may induce synergistic anti-cancer activity and immune responses in pancreatic cancer. Effective harnessing of the immune system and rational combinations with stroma-targeting biological agents (PEGPH20) is a novel field that needs to be explored in pancreatic cancer. This phase II trial will determine the efficacy of pembrolizumab plus PEGPH20 in metastatic pancreatic cancer patients who have HA-high tumor expression. Stroma and immune-related biomarkers will be tested prospectively in blood and tumor biopsies at baseline, after 6 weeks of therapy, and at time of cancer progression. A phase I study with pembrolizumab and PEGPH20 is ongoing in lung and gastric cancer patients (NCT02563548), and demonstrated safety and tolerability of this combination at the doses administered in this study (Halozyme data).

Immunotherapies have the potential to induce durable therapeutic responses although this typically occurs in a small fraction of patients. Biomarker-guided patient selection can, in principle, identify those patients most likely to benefit. The investigators hypothesize that stroma remodeling with PEGPH20 will potentiate effector CD8 T cell lymphocyte infiltration and sensitize pancreatic cancer to immune therapy, and that immunologic, and/or genomic biomarkers will identify patient subsets most likely to benefit. As examples, MSI-high status and high tumor mutational burden (hypermutation) have been linked to sensitivity to immune checkpoint inhibitors (Le et al. 2015, Le et al. 2016).

Assays may include but are not limited to: Immunohistochemical analysis, profiling of the immune transcriptome, circulating cytokine analyses, flow cytometric analyses of peripheral and intratumoral immune response.

This is an open label non-randomized Phase II trial for patients with previously treated metastatic ductal pancreatic adenocarcinoma with HA-high expression, to assess the progression-free survival rate (PFS) of patients treated with this combination therapy. Secondary endpoints will assess safety and tolerability, overall response rate (ORR), disease control rate (DCR= CR+PR+SD), duration of response and stable disease (DOR), and overall survival (OS).

There will be an estimated 35 patients enrolled into the study, using 5 centers in the U.S.

Overall response rates as well as individual categories of response (CR, PR, SD, and PD) will be determined using RECIST 1.1. Time-to-event endpoints, including PFS and OS will be assessed using the Kaplan-Meier method. Toxicity (adverse events) will be recorded using the NCI CTCAE, version 5.0 (published Nov 2017, Appendix B).

All patients will start treatment with PEGPH20 3 microgram/kg IV weekly x 3, and pembrolizumab 200 mg IV every 3 weeks, in 3-week cycles.

Patients may remain on treatment with PEGPH20 in combination with pembrolizumab as long as they are receiving clinical benefit, until disease progression per RECIST 1.1 criteria, or until untolerable toxicity develops, whichever comes first. If no disease progression, patients will be allowed to remain on study treatment for up to 24 months. If no disease progression, but with unacceptable toxicity from PEGPH20, patients will be allowed to continue on pembrolizumab alone for up to 24 months if deemed appropriate by the investigator. If pembrolizumab needs to be discontinued for toxicity, patients may continue treatment with PEGPH20 alone.

The estimated duration for accrual is anticipated to be 12 months. Patients will be followed up for a minimum of 6 months. The overall study duration is estimated at approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Histologically confirmed metastatic pancreatic ductal adenocarcinoma, via archived or fresh core biopsy of either primary tumor or metastatic site.
3. Available tumor tissue (formalin-fixed paraffin-embedded [FFPE] block preferred) with enough tumor to make a minimum of 5-10 unstained, consecutive FFPE slides (10 slides are preferred) of 1 archival block that meets specific tissue sample requirements. Archived or fresh tissue from the primary lesion or a metastatic lesion is required. Note: Fine needle aspirates or brushing biopsies will not be acceptable. This tumor tissue requirement is for the determination of the HA-high or -low expression status.
4. Subjects must be determined to be HA-high based on archival or fresh tumor biopsy that meets the requirements noted in the previous inclusion criterion.
5. 18 years of age on day of signing informed consent.
6. Have measurable metastatic disease based on RECIST 1.1.
7. Life expectancy ≥ 12 weeks.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Received no more than 2 prior lines of systemic therapy for metastatic disease (1 or 2 prior lines of therapy for metastatic disease are allowed)
10. Be willing to provide tumor tissue from newly obtained tumor cores or excisional biopsy for research purposes. Newly-obtained is defined as a specimen obtained within 2 weeks (14 days) prior to initiation of treatment on Day 1.
11. Be willing to provide tumor tissue from tumor biopsy after 6 weeks of treatment (mandatory, if safe and feasible), and at the time of tumor progression (optional, if safe and feasible). Note: Fine needle aspirates or brushing biopsies will not be acceptable.
12. Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation.
13. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
16. No history of acute DVT/PE or CVA/TIA (new within 4 weeks of study registration) or clinical significant carotid artery disease.
17. If prior history of DVT/PE the patient needs to be on stable doses of anticoagulation with low molecular weight heparins.

    * Patients should have all eligibility criteria met, before undergoing the baseline research biopsy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (equivalent of > 20 mg of hydrocortisone per day) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active tuberculosis (TB).
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Known allergy to PEGPH20 (hyaluronidase).
6. Current use of megestrol acetate (use within 10 days of Day 1).
7. Contraindication to heparin as per institutional guidelines.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier.
9. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs), or documented history of clinically severe autoimmune disease (e.g., colitis, Crohns' disease)*. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

    *Any relevant diseases that are not listed as examples of exclusionary diseases are to be discussed with the Sponsor-Investigator.
13. Has known history of, or any evidence of active, non-infectious pneumonitis.
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
15. Has known hepatobiliary diseases (e.g., primary biliary cholangitis, primary sclerosing cholangitis, immune mediated cholangitis); patients with cholangitis attributed to infectious etiology (e.g., ascending cholangitis, bacterial cholangitis) are eligible if the infection has been fully recovered prior to the screening visit.
16. Has known history of drug-induced hepatobiliary toxicities
17. Has an active infection requiring systemic therapy.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
21. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or any other immune checkpoint inhibitors.
22. Has received prior therapy with PEGPH20, or has participated in the Halozyme HALO 301 phase III study.
23. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
24. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
25. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | PFS will be assessed from Date of registration through study closure, up to 24 months. PFS is calculated as the number of days from date of registration to date of disease progression or symptomatic deterioration, or death due to any cause.
  Evaluate the progression-free survival (PFS) for patients treated with pembrolizumab and PEGPH20

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Safety and Tolerability using CTCAE v5.0 will be assessed from Day 1 of study treatment through 30-days past the last study treatment per patient, through study closure, up to 24 months.
  Evaluate the safety and tolerability of this treatment combination as assessed by CTCAE v5.0.
Overall Response Rate | ORR is assessed from Day 1 of treatment to study closure, up to 24 months. ORR is calculated by adding the Complete Responses (CR) with the Partial Responses (PR), based on RECIST v1.1, recorded at each disease evaluation for each patient.
  Evaluate the Overall Response Rate (ORR, CR + PR) based on RECIST v1.1
Disease Control Rate | DCR is assessed from Day 1 of treatment to study closure, up to 24 months. DCR is calculated by adding the Complete Responses, Partial Responses and Stable Disease, based on RECIST v1.1, recorded at each disease evaluation for each patient.
  Evaluate Disease Control Rate (DCR, CR +PR+SD)
Duration of Response | DOR is assessed from Day 1 of treatment to study closure, up to 24 months. DOR is calculated for patients who achieve a CR or PR, as the number of days from the date of response to the date of progression, or death, due to any cause.
  Evaluate the Duration of Response (DOR)
Overall Survival | Overall Survival is assessed from date of registration to study closure, up to 24 months. Overall Survival is calculated as the number of days from date of registration to date of death due to any cause.
  Evaluate the Overall Survival

OTHER OUTCOMES:
Evaluate Plasma Hyaluronan (HA) levels | Plasma Hyaluronan (HA) levels are measured in blood samples taken at Day 1 of every treatment cycle (1 cycle = 3 weeks), during each patient's study treatment, with data from these samples assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatments plasma hyaluronan (HA) levels in blood samples, and correlate with ORR, PFS, and OS
Evaluate immunological biomarkers using flow cytometry in tumor tissue samples | Immunological biomarkers using flow cytometry are measured in tumor tissue samples taken at 3 timepoints during each patient's study treatment, with data from these samples assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment immunological biomarkers (the percentage and absolute count (cells/mm3) of T-cell subsets) using flow cytometry, in tumor tissue samples and correlate with ORR, PFS, and OS
Evaluate immunological biomarkers--T-cell receptor (TCR) sequencing in tumor tissue samples | Immunological biomarkers of T-cell receptor (TCR) sequencing are measured in tumor tissue samples taken at 3 timepoints during each patient's study treatment, with data from these samples assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment immunological biomarkers of T-cell receptor (TCR) sequencing in tumor tissue samples, and correlate with ORR, PFS, and OS
Evaluate immunological biomarkers--focused gene profiling of the immune transcriptome | Immunological biomarkers--focused gene profiling of the immune transcriptome--are measured in tumor tissue samples taken at 3 timepoints during each patient's study treatment, with data assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment immunological biomarkers--focused gene profiling of the immune transriptome--in tumor tissue samples, and correlate with ORR, PFS, and OS
Evaluate immunological biomarkers--Immunohistochemistry (IHC) for T-cells, B-cells, and macrophages subsets | Immunological biomarkers--IHC of T-cells, B-cells and macrophages subsets are measured in tumor tissue samples taken at 3 timepoints during each patient's study treatment, with data assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment immunological biomarkers--IHC of T-cells, B-cells, and macrophages subsets-- in tumor tissue samples, and correlate with ORR, PFS, and OS
Evaluate Blood Translational Biomarker--Circulating cytokines/chemokines in plasma | The Translational Biomarkers-- circulating cytokines/chemokines in plasma-- are measured in blood samples taken at 3 timepoints during each patient's study treatment, with data from these samples assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment Translational biomarkers of circulating cytokines/chemokines in plasma blood samples and correlate with ORR, PFS, and OS
Evaluate Blood Translational Biomarkers--flow cytometry | The Translational Biomarkers using flow cytometry are measured in blood samples taken at 3 timepoints during each patient's study treatment, with data assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment Translational biomarkers in blood samples (the percentage and absolute count (cells/mm3) of T-cell subsets) using flow cytometry, and correlate with ORR, PFS, and OS
Evaluate Blood Translational Biomarkers--T cell receptor (TCR) sequencing | The Translational Biomarker-- T-cell receptor (TCR) sequencing-- are measured in blood samples taken at 3 timepoints during each patient's study treatment, with data from these samples assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment Translational biomarkers of T-cell receptor (TCR) sequencing in blood samples and correlate with ORR, PFS, and OS

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Chiorean, MD, Principal Investigator — Seattle Cancer Care Alliance--University of Washington
Locations (5):
- United States (5):
  - Banner Health - MD Anderson Cancer Center, Gilbert, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rutgers - Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey
  - University of Washington--Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] 46. Le DT, Uram JN, Wang H, et al. PD-1 blockade in mismatch repair deficient non-colorectal gastrointestinal cancers. J Clin Oncol . 2016. 34 (suppl 4S; abstr 195).